CLINICAL TRIAL: NCT01942070
Title: Intracoronary Scaffold Assessment a Randomised Evaluation of Absorb in Myocardial Infarction (ISAR-Absorb MI) A Prospective, Randomized Trial of BVS Veruss EES in Patients Undergoing Coronary Stenting for Myocardial Infarction
Brief Title: A Prospective, Randomized Trial of BVS Veruss EES in Patients Undergoing Coronary Stenting for Myocardial Infarction
Acronym: ISAR-Absorb MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ge IDE No. I01210
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Cardiovascular Disease; Myocardial Infarction; Thrombus; Primary Angioplasty
Keywords: Cardiovascular Disease; Myocardial Infarction; Bioresorbable vascular scaffold; Durable polymer everolimus-eluting stent; Primary angioplasty; Stent
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bioresorbable vascular scaffold (Experimental): Bioresorbable vascular scaffold (BVS)
  Interventions: Device: Bioresorbable vascular scaffold
- Everolimus-eluting stent (Active Comparator): Durable polymer everolimus-eluting metallic stent (EES)
  Interventions: Device: Durable polymer everolimus-eluting metallic stent

INTERVENTIONS:
Device: Bioresorbable vascular scaffold
  Other Names: ABSORB
  Arms: Bioresorbable vascular scaffold
Device: Durable polymer everolimus-eluting metallic stent
  Other Names: Xience
  Arms: Everolimus-eluting stent

SUMMARY:
The aim of the current study is to test the clinical performance of the everolimus-eluting BVS compared with that of the durable polymer everolimus-eluting stent (EES) in patients undergoing PCI in the setting of acute MI.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) with drug-eluting stent (DES) implantation currently represents the dominant treatment strategy in patients undergoing catheter intervention. However effective neointimal suppression occurs at the cost of a systematic delay in arterial healing in comparison with after bare metal stenting. This underlies a small but significant increased risk of stent thrombosis after DES implantation in comparison with bare metal stent implantation as well as a possible excess of in-stent neoatheroma formation.

Bioresorbable vascular scaffolds (BVS) represent an innovative technology providing short-term vessel scaffolding and drug delivery without the long-term limitations of metallic DES and durable polymer coatings. Potential benefits include restoration of normal vasomotor reactivity, facilitation of positive vessel wall remodelling and facilitation of subsequent bypass grafting of the stented arterial segment. In addition preliminary reports suggest that the process of scaffold biodegradation may promote formation of a cohesive tissue layer covering and stabilizing the underlying atherosclerotic plaque - a so-called plaque-sealing effect. Although initial results with BVS are encouraging, there is a lack of randomized clinical trial data and no data exists for outcomes after BVS implantation in patients undergoing coronary stenting in the setting of acute myocardial infarction (MI).

The aim of the current study is to test the clinical performance of the everolimus-eluting BVS compared with that of the durable polymer everolimus-eluting stent (EES) in patients undergoing PCI in the setting of acute MI. The primary endpoint will be percentage diameter stenosis at protocol-mandated 6-8 month angiographic follow-up. Sample size calculation is based on a non-inferiority assumption in relation to the BVS versus EES. It is planned to enrol a total of 260 patients. Subsequent clinical follow-up will be undertaken out to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older with acute ST-elevation myocardial infarction or non ST-elevation myocardial infarction with angiographically confirmed thrombus
2. Planned stent implantation in de novo lesions in native vessels or coronary bypass grafts with reference vessel diameter ≥2.5 mm and ≤3.9 mm
3. Written, informed consent by the patient or her/his legally-authorized representative for participation in the study
4. In women with childbearing potential a negative pregnancy test is mandatory

Exclusion Criteria:

1. Target lesion located in the left main trunk
2. Severely calcified lesions
3. Bifurcation lesions with side branch diameter > 2mm
4. In-stent restenosis
5. Contraindications to antiplatelet therapy, cobalt chrome, everolimus, polylactic acid
6. Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance
7. Pregnancy (present, suspected or planned) or positive pregnancy test.
8. Previous enrolment in this trial
9. Patient's inability to fully cooperate with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Percentage Diameter Stenosis | 6-8 months
  Percentage diameter stenosis at coronary angiography at 6-8 months follow-up

SECONDARY OUTCOMES:
Device-oriented composite endpoint | 12 months
  Composite of cardiac death/target vessel-myocardial infarction (MI)/ target lesion revascularization (TLR)
Patient-oriented composite endpoint | 12 months
  The composite of death/any MI/all revascularization
Composite of death or MI | 12 months
  The composite of cardiovascular death or MI
Stent thrombosis | 12 months
  The incidence of scaffold or stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Byrne, MB PhD, Principal Investigator — Deutsches Herzzentrum Munich
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Munich, Munich, Bavaria
  - Klinikum Rechts der Isar, Munich, Bavaria

REFERENCES:
- [Derived] Cassese S, Katagiri Y, Byrne RA, Brugaletta S, Alfonso F, Raber L, Maeng M, Iniguez A, Kretov E, Onuma Y, Joner M, Sabate M, Laugwitz KL, Windecker S, Kastrati A, Serruys PW. Angiographic and clinical outcomes of STEMI patients treated with bioresorbable or metallic everolimus-eluting stents: a pooled analysis of individual patient data. EuroIntervention. 2020 Mar 20;15(16):1451-1457. doi: 10.4244/EIJ-D-18-01080. PMID 30719976
- [Derived] Byrne RA, Alfonso F, Schneider S, Maeng M, Wiebe J, Kretov E, Bradaric C, Rai H, Cuesta J, Rivero F, Hoppmann P, Schlichtenmaier J, Christiansen EH, Cassese S, Joner M, Schunkert H, Laugwitz KL, Kastrati A. Prospective, randomized trial of bioresorbable scaffolds vs. everolimus-eluting stents in patients undergoing coronary stenting for myocardial infarction: the Intracoronary Scaffold Assessment a Randomized evaluation of Absorb in Myocardial Infarction (ISAR-Absorb MI) trial. Eur Heart J. 2019 Jan 7;40(2):167-176. doi: 10.1093/eurheartj/ehy710. PMID 30520980